CLINICAL TRIAL: NCT01339923
Title: A Phase 3B, Open Label, Multi-Center Study to Evaluate the Safety, Tolerability and Immunogenicity of Novartis Meningococcal B Recombinant Vaccine When Administered Alone to Healthy Infants According to Different Immunization Schedules and to Healthy Children Aged 2 to 10 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V72_28
Record Dates: First submitted 2011-04-13; First posted 2011-04-21 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-03

CONDITIONS: Meningococcal Disease; Meningococcal Meningitis
Keywords: Meningococcal disease; Vaccines; intercalated administration
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- B_2h3h5_11 (Experimental): Subjects, approximately 2.5 months of age, received 3 dose primary vaccination of rMenB+OMV NZ at 2.5, 3.5, 5 months of age, followed by a booster dose at 11 months of age.
  Interventions: Biological: rMenB + OMV NZ vaccine
- B_3h5_11 (Experimental): Subjects, approximately 3.5 months of age, received 2 dose primary vaccination of rMenB+OMV NZ at 3.5 and 5 months of age, followed by a booster dose at 11 months of age.
  Interventions: Biological: rMenB + OMV NZ vaccine
- B_68_11 (Experimental): Subjects, approximately 6 months of age, received 2 dose primary vaccination of rMenB+OMV NZ at 6 and 8 months of age, followed by a booster dose at 11 months of age.
  Interventions: Biological: rMenB + OMV NZ vaccine
- B_02_2_5 (Experimental): Subjects, 2-5 years of age received 2 catch-up doses of rMenB+OMV NZ, each at 0 and 2 months. Blood draw at 0 and 3 months since study start.
  Interventions: Biological: rMenB + OMV NZ vaccine
- B_02_6_10 (Experimental): Subjects, 6-10 years of age received 2 catch-up doses of rMenB+OMV NZ, each at 0 and 2 months. Blood draw at 0 and 3 months since study start.
  Interventions: Biological: rMenB + OMV NZ vaccine
- BC_35_12 (Experimental): Subjects, 3 months of age received rMenB+OMV NZ + MenC-CRM and Synflorix concomitantly at 3, 5 and 12 months of age and an additional dose of Synflorix alone dose at 7 months of age.
  Interventions: Biological: Meningococcal C oligosaccharide conjugated vaccine; Biological: Pneumococcal polysaccharide conjugate vaccine, 10 valent adsorbed.; Biological: rMenB + OMV NZ vaccine
- C_35_12 (Experimental): Subjects, 3 months of age received MenC-CRM and Synflorix concomitantly at 3, 5 and 12 months of age and an additional dose of Synflorix alone at 7 months of age and rMenB+OMV NZ alone at 13 and 15 months of age.
  Interventions: Biological: Meningococcal C oligosaccharide conjugated vaccine; Biological: Pneumococcal polysaccharide conjugate vaccine, 10 valent adsorbed.; Biological: rMenB + OMV NZ vaccine

INTERVENTIONS:
Biological: rMenB + OMV NZ vaccine — 3 doses (2.5, 3.5, 5 months if age) plus booster (11 months of age)
  Other Names: rMenB for Group I
  Arms: B_2h3h5_11
Biological: rMenB + OMV NZ vaccine — 2 doses (3.5, 5 months of age) plus booster (11 months of age)
  Other Names: rMenB for Group II
  Arms: B_3h5_11
Biological: rMenB + OMV NZ vaccine — 2 doses (6, 8 months of age) plus booster (11 months of age)
  Other Names: rMenB for Group III
  Arms: B_68_11
Biological: rMenB + OMV NZ vaccine — 2 doses 2 months apart
  Other Names: rMenB for Group IV
  Arms: B_02_2_5; B_02_6_10
Biological: Meningococcal C oligosaccharide conjugated vaccine — Schedule 3, 5, 7, 12, Meningococcal C oligosaccharide conjugated vaccine
  Arms: BC_35_12; C_35_12
Biological: Pneumococcal polysaccharide conjugate vaccine, 10 valent adsorbed. — Schedule 3, 5, 7, 12 Pneumococcal polysaccharide conjugate vaccine, 10 valent adsorbed.
  Arms: BC_35_12; C_35_12
Biological: rMenB + OMV NZ vaccine — Schedule 3, 5, 12 rMenB + OMV vaccine
  Other Names: rMenB for Group V
  Arms: BC_35_12
Biological: rMenB + OMV NZ vaccine — Schedule 13,15 rMenB + OMV vaccine
  Other Names: rMenB for Group VI
  Arms: C_35_12

SUMMARY:
The proposed study is aimed at assessing the safety and immunogenicity of rMenB+OMV NZ when administered alone without routine infant vaccines to healthy infants in their first year of life according to different two and three dose immunization schedules, which are suitable to be adopted by various national programs. This study will also investigate antibody persistence post primary series and administration of a subsequent booster dose of rMenB+OMV NZ at 11 months of age. In addition, this study will assess the safety and immunogenicity of two catch-up doses of rMenB+OMV NZ when administered to healthy children 2 to 10 years of age.

This study will also evaluate the safety and immunogenicity of the concomitant administration of rMenB+OMV NZ with meningococcal C conjugate vaccine (MenC-CRM) according to a 3, 5 and 12-month schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants and children according to the following age groups:

   * Healthy infants 2½ months of age (71 -79 days, inclusive), (only applicable to group I)
   * Healthy infants 3½ months of age (101 -109 days, inclusive), (only applicable to group II)
   * Healthy infants 6 months of age (only applicable to group III) (The age window is defined as the first day the subject turns 6 months of age up to the day before the subject turns 7 months of age).
   * Healthy children 2 to 5 years of age (only applicable to group IVa) (The age window is defined as the first day the subject turns 2 years of age up to the day before the subject turns 6 years of age).
   * Healthy children 6 to 10 years of age (only applicable to group IVb) (The age window is defined as the first day the subject turns 6 years of age up to the day before the subject turns 11 years of age).
   * Healthy infants 3 months of age (83-104 days, inclusive), (only applicable to Group V and VI).
2. For whom parent(s)/legal guardian(s) have given written informed consent according to local regulations after the nature of the study has been explained;
3. Available for all the visits scheduled in the study;
4. Individuals in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator.

Exclusion Criteria:

1. Individuals whose parent(s)/legal guardian(s) are unwilling or unable to give written informed consent to participate in the study;
2. Children's parents or legal guardian who are not able to comprehend and to follow all required study procedures for the whole period of the study.
3. History of any meningococcal B vaccine administration;
4. Previous ascertained or suspected disease caused by N. meningitidis;
5. Household contact with and/or intimate exposure to an individual with laboratory confirmed N. meningitidis;
6. History of severe allergic reaction after previous vaccinations or hypersensitivity to any vaccine component
7. Significant acute or chronic infection within the previous 7 days or temperature 38° C within the previous day of receiving the study vaccine;
8. Antibiotics treatment within 6 days prior to enrollment;
9. Individuals with history of allergy to vaccine components.
10. Any serious chronic or progressive disease according to the judgment of the investigator (e.g., neoplasm, diabetes mellitus Type I, cardiac disease, hepatic disease, neurological disease or seizure, either associated with fever or as part of an underlying neurological disorder or syndrome, autoimmune disease, HIV infection or AIDS, or blood dyscrasias or diathesis, signs of cardiac or renal failure or severe malnutrition);
11. Known or suspected impairment/alteration of the immune system, immunosuppressive therapy, use of high dose systemic corticosteroids or chronic use of inhaled high-potency corticosteroids within 14 days prior to enrollment (use of low or moderate doses of inhaled steroids is not an exclusion);
12. Receipt of blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation within 90 days prior to enrollment.
13. Receipt of, or intent to immunize with, any other vaccine(s) within 7 days prior to enrollment.
14. Individuals participating in any clinical trial with another investigational product 30 days prior to first study visit or intent to participate in another clinical study at any time during the conduct of this study.
15. Family members and household members of research staff
16. Individuals with history or any illness that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study.
17. History of any meningococcal C vaccine administration (Only applicable to group V and VI).
18. History of any Pneumococcal vaccine administration (Only applicable to group V and VI).

Ages: 71 Days to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1409 (Actual)
Dates: Start 2011-04; Primary Completion 2014-01 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (26):
- Brazil (4):
  - Site 55 - Instituto de Medicina Integral Prof. Fernando Figueira (IMIP), Rua Dos Coelhos, 300 - Boa Vista, Recife/PE
  - Site 54- Associação Obras Sociais Irmã Dulce, Avenida Bonfim, nº 161, Largo de Roma, Salvador/BA-CEP
  - Site 53 - CRIE UNIFESP, Rua Borges Lagoa 770, São Paulo
  - Site 50 - Associacao Fundo de Incentivo a Psicofarmacologia, Rua Marselhesa 500 Vila Clementino, São Paulo
- Hungary (10):
  - Site 37 - Praxis Dr Julianna Kovacs, Honved Utca 2, Bordany
  - Site 40 - General Pediatric Practice Hacsek, Poth Iren U 80, Budapest
  - Site 42 - Praxis Dr Eszter Bari, Szentharomsag Ter 10, Csongrád megye
  - Site 34 - General Pediatric Practice Somorjai, Bajcsi Ut 32, Debrecen
  - Site 32 - Praxis Dr Eleonora Konya, Fo Utca 12, Malyi
  - Site 31 - General Practice Dr Olga Fekete, Kando Kalman Utca 1, Miskolc
  - Site 30 - General Practice Dr Simko, Selyemret U. 1., Miskolc
  - Site 33 - General Pediatric Practice Ujhelyi, Szent Istvan U 10, Nyiregyhaza
  - Site 35 - Praxis Dr Eva Kovacs, Csongradi Sgt 63, Szeged
  - Site 36 - General Practice Dr Edit Oszlacs, Debreceni Utca 10-14, Szeged
- Peru (3):
  - Site 80 - Hospital Nacional docente Madre Nino San Bartolome, Av Alfonso Ugarte, Lima
  - Site 82 - Investigaciones Medicas en Salud INMENSA, Jr Jose de La Torre Ugarte Lince, Lima
  - Site 81 - Via Libre, Jr Paraguay Cercado de Lima, Lima
- Spain (9):
  - Site 15, Almería
  - Site 16, Almería
  - Site 20, Barcelona
  - Site 17, Madrid
  - Site 18, Madrid
  - Site 11, Ourense
  - Site 13, Pontevedra
  - Site 10, Santiago de Compostela
  - Site 14, Seville

REFERENCES:
- [Derived] Safadi MAP, Martinon-Torres F, Weckx LY, Moreira ED Junior, da Fonseca Lima EJ, Willemsen A, Toneatto D, Habib MA, Borys D. Immunogenicity of the pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) administered concomitantly with the meningococcal serogroup B (4CMenB) vaccine in infants: A post-hoc analysis in a phase 3b, randomised, controlled trial. Vaccine. 2019 Aug 14;37(35):4858-4863. doi: 10.1016/j.vaccine.2019.07.021. Epub 2019 Jul 18. PMID 31327652
- [Derived] Martinon-Torres F, Carmona Martinez A, Simko R, Infante Marquez P, Arimany JL, Gimenez-Sanchez F, Couceiro Gianzo JA, Kovacs E, Rojo P, Wang H, Bhusal C, Toneatto D. Antibody persistence and booster responses 24-36 months after different 4CMenB vaccination schedules in infants and children: A randomised trial. J Infect. 2018 Mar;76(3):258-269. doi: 10.1016/j.jinf.2017.12.005. Epub 2017 Dec 15. PMID 29253560
- [Derived] P Safadi MA, Martinon-Torres F, Weckx LY, Moreira ED Junior, da Fonseca Lima EJ, Mensi I, Calabresi M, Toneatto D. Immunogenicity and safety of concomitant administration of meningococcal serogroup B (4CMenB) and serogroup C (MenC-CRM) vaccines in infants: A phase 3b, randomized controlled trial. Vaccine. 2017 Apr 11;35(16):2052-2059. doi: 10.1016/j.vaccine.2017.03.002. Epub 2017 Mar 18. PMID 28318767

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in a total of a total of 26 sites; 4 sites in Brazil, 3 sites in Peru, 10 sites in Hungary, 9 sites in Spain.
Pre-assignment Details: All enrolled subjects were included in the study.
Groups:
- B_2h3h5_11: Subjects, approximately 2.5 months of age received 3 dose primary vaccination of rMenB+OMV NZ at 2.5, 3.5, 5 months of age, followed by a booster dose at 11 months of age.
- B_3h5_11: Subjects, approximately 3.5 months of age received 2 dose primary vaccination of rMenB+OMV NZ at 3.5 and 5 months of age, followed by a booster dose at 11 months of age.
- B_68_11: Subjects, approximately 6 months of age received 2 dose primary vaccination of rMenB+OMV NZ at 6 and 8 months of age, followed by a booster dose at 11 months of age.
Period: Overall Study
Arm/Group | B_2h3h5_11 | B_3h5_11 | B_68_11 | B_02_2_5 | B_02_6_10 | BC_35_12 | C_35_12
Started | 253 | 250 | 251 | 104 | 300 | 126 | 125
Completed | 239 | 234 | 243 | 100 | 295 | 117 | 111
Not Completed | 14 | 16 | 8 | 4 | 5 | 9 | 14
Not completed — Adverse Event | 1 | 1 | 1 | 0 | 0 | 0 | 1
Not completed — Inappropriate Enrollment | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 4 | 4 | 0 | 3 | 1 | 1 | 5
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 3 | 1
Not completed — Unable to Classify | 1 | 0 | 1 | 0 | 0 | 1 | 5
Not completed — Withdrawal by Subject | 7 | 11 | 6 | 1 | 4 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- TOTAL: Total of all reporting groups
Arm/Group | B_2h3h5_11 | B_3h5_11 | B_68_11 | B_02_2_5 | B_02_6_10 | BC_35_12 | C_35_12 | TOTAL
Number analyzed (Participants) | 253 | 250 | 251 | 104 | 300 | 126 | 125 | 1409
Age, Continuous [Mean (Standard Deviation); unit: month] | 2.0 (0.1) | 3.0 (0.1) | 6.0 (0.0) | 47.5 (13.4) | 96.9 (16.8) | 3.0 (0.2) | 3.0 (0.1) | 26.6 (39.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 124 | 127 | 49 | 149 | 74 | 59 | 699
  Male | 136 | 126 | 124 | 55 | 151 | 52 | 66 | 710

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With Serum Bactericidal Activity Using Human Serum (hSBA) Titers ≥ 4 or hSBA Titers ≥ 5 (Strain M10713) Following a 2-dose Primary Series of rMenB+OMV Vaccination.
Description: Immunogenicity was assessed in terms of percentages of subjects with hSBA titers ≥ 4 against N meningitidis serogroup B strains H44/76, 5/99, NZ98/254 and hSBA titers ≥ 5 against strain M10713 following 2-dose primary series of vaccination with rMenB+OMV NZ at 3.5 and 5 months of age or at 6 and 8 months of age. Analysis was done on Full analysis set (FAS)-Primary series.
Time Frame: 1 month after second vaccination
Population: FAS-Primary series
Measure: Number (97.5% Confidence Interval); unit: Percentages of subjects
Arm/Group | B_3h5_11 | B_68_11
Number analyzed (Participants) | 230 | 238
Percentages of subjects
  H44/76 (hSBA≥ 4; N=228, 234)) | 100 [97 to 100] | 100 [97 to 100]
  5/99 (hSBA≥ 4) | 100 [97 to 100] | 100 [98 to 100]
  NZ98/254 (hSBA≥ 4; N=230, 233) | 98 [95 to 99] | 99 [97 to 100]
  M10713 (hSBA≥ 5; N=181, 192)) | 44 [35 to 52] | 73 [65 to 80]

2. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 4, hSBA Titers ≥ 5 (Strain M10713) and hSBA ≥ 8 Following a 3-dose Primary Series of rMenB+OMV Vaccination
Description: Immunogenicity was assessed in terms of percentages of subjects with hSBA titers ≥ 4 against N meningitidis serogroup B strains H44/76, 5/99, NZ98/254; hSBA titers ≥ 5 against strain M10713 and hSBA titers ≥ 8 against strains H44/76, 5/99, NZ98/254, M10713, following 3-dose primary series of vaccination with rMenB+OMV NZ at 2.5, 3.5 and 5 months of age. Analysis was done on FAS-primary series.
Time Frame: 1 month after third vaccination
Population: FAS-primary series
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- B_2h3h5_11: Subjects, approximately 2.5 months of age, received 3 dose primary vaccination of rMenB+OMV NZ at 2.5, 3.5, 5 months of age, followed by a booster dose at 11 months of age.
  rMenB + OMV NZ vaccine: 3 doses (2.5, 3.5, 5 months of age) plus booster (11 months of age)
Arm/Group | B_2h3h5_11
Number analyzed (Participants) | 238
Percentages of subjects
  H44/76 (hSBA≥ 4; 1 month after 3rd vacc; N=237) | 100 [98 to 100]
  5/99 (hSBA≥ 4; 1 month after 3rd vacc) | 100 [98 to 100]
  NZ98/254 (hSBA≥ 4; 1 month after 3rd vacc) | 99 [96 to 100]
  M10713 (hSBA≥ 5; 1 month after 3rd vacc; N=197) | 55 [48 to 62]
  H44/76 (hSBA≥ 8; 1 month after 3rd vacc; N=237) | 98 [96 to 100]
  5/99 (hSBA≥ 8; 1 month after 3rd vacc) | 100 [98 to 100]
  NZ98/254 (hSBA≥ 8; 1 month after 3rd vacc) | 89 [85 to 93]
  M10713 (hSBA≥ 8; 1 month after 3rd vacc; N=197) | 47 [40 to 54]

3. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 4 or hSBA Titers ≥ 5 (Strain M10713) and hSBA ≥ 8 Following a 2-dose Catch-up Series of rMenB+OMV Vaccination
Description: Immunogenicity was assessed in terms of percentages of subjects with hSBA titers ≥ 4 against N meningitidis serogroup B strains H44/76, 5/99, NZ98/254; hSBA titers ≥ 5 against strain M10713 and hSBA titers ≥ 8 against strains H44/76, 5/99, NZ98/254, M10713; following 2-dose catch-up series of vaccination with rMenB+OMV NZ in healthy children aged 2-10 years (0, 2 month schedule). Analysis was done on FAS-primary series.
Time Frame: 1 month after second vaccination
Population: FAS-primary series
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- B_02: Subjects, 2-10 years of age received 2 catch-up doses of rMenB+OMV NZ, each at 0 and 2 months. Blood draw at 0 and 3 months since study start.
  rMenB + OMV NZ vaccine: 2 doses 2 months apart
Arm/Group | B_02
Number analyzed (Participants) | 390
Percentages of subjects
  H44/76 (hSBA≥ 4; 1 month after 2nd vacc; N=386) | 99 [97 to 100]
  5/99 (hSBA≥ 4; 1 month after 2nd vacc) | 99 [98 to 100]
  NZ98/254 (hSBA≥ 4; 1 month after 2nd vacc; N=389) | 99 [97 to 100]
  M10713 (hSBA≥ 5; 1 month after 2nd vacc; N=370) | 94 [91 to 96]
  H44/76 (hSBA≥ 8; 1 month after 2nd vacc; N=386) | 98 [96 to 99]
  5/99 (hSBA≥ 8; 1 month after 2nd vacc) | 99 [98 to 100]
  NZ98/254 (hSBA≥ 8; 1 month after 2nd vacc; N=389) | 95 [92 to 97]
  M10713 (hSBA≥ 8; 1 month after 2nd vacc; N=370) | 92 [89 to 94]

4. Secondary Outcome: Percentages of Subjects Achieving Four-fold Rise Over Baseline hSBA Titers Following a 2-dose Catch-up Series of rMenB+OMV Vaccination
Description: Immunogenicity was assessed in terms of percentages of subjects achieving 4-fold increase in hSBA titers as compared to baseline against N meningitidis serogroup B strains H44/76, 5/99, NZ98/254, M10713; following 2-dose catch-up series of vaccination with rMenB+OMV NZ in healthy children aged 2-10 years (0, 2 month schedule).
  Analysis was done on FAS- primary series.
Time Frame: 1 month after second vaccination
Population: FAS- primary series
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | B_02
Number analyzed (Participants) | 388
Percentages of subjects
  H44/76 (1 month after 2nd vacc; N=385) | 96 [93 to 97]
  5/99 (1 month after 2nd vacc) | 99 [97 to 100]
  NZ98/254 (1 month after 2nd vacc; N=387) | 93 [89 to 95]
  M10713 (1 month after 2nd vacc; N=352) | 46 [41 to 51]

5. Secondary Outcome: Geometric Mean hSBA Titers (GMTs) Following 2 or 3 Dose Primary Series of Vaccination With rMenB+OMV
Description: Immunogenicity was assessed in terms of Geometric mean hSBA titers (GMTs) against N meningitidis serogroup B indicator strains following 2 or 3 dose primary series of vaccination rMenB+OMV NZ (1 month after 3rd infant vaccination in B_2h3h5_11 and 1 month after 2nd infant vaccination in B_3h5_11, B_68_11 and B_02).
  Analysis was done on FAS-primary series.
Time Frame: 1 month after primary series vaccination
Population: FAS-primary series
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | B_2h3h5_11 | B_3h5_11 | B_68_11 | B_02
Number analyzed (Participants) | 238 | 230 | 238 | 390
Titers
  H44/76 (1 month after primary vacc; N=237,228,234, | 109 [92 to 130] | 132 [110 to 158] | 240 [201 to 287] | 121 [109 to 135]
  5/99 (1 month after primary vacc) | 795 [665 to 950] | 605 [502 to 729] | 1157 [964 to 1390] | 489 [442 to 541]
  NZ98/254 1m after primary vacc; N=238,230,233,389 | 34 [28 to 42] | 39 [31 to 48] | 65 [52 to 80] | 42 [38 to 47]
  M10713 1 m after primary vacc; N=197,181,192,370 | 4.86 [3.62 to 6.54] | 3.39 [2.48 to 4.64] | 9.96 [7.33 to 14] | 35 [31 to 39]

6. Secondary Outcome: Geometric Mean hSBA Titers (GMTs) After First Infant Vaccination With rMenB+OMV.
Description: Immunogenicity was assessed in terms of Geometric mean hSBA titers (GMTs) against N meningitidis serogroup B indicator strains after the first infant vaccination in groups B_2h3h5_11b, B_3h5_11b and B_68_11b (after 1 month for group B_2h3h5_11b, 1.5 months for group B_2h3h5_11b and 2 months for group B_68_11b). Analysis was done on FAS-post first dose.
Time Frame: 1, 1.5 or 2 months after first infant vaccination
Population: FAS-post first dose
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- B_2h3h5_11b: Subjects, approximately 2.5 months of age, received 3 dose primary vaccination of rMenB+OMV NZ at 2.5, 3.5, 5 months of age, followed by a booster dose at 11 months of age. Blood draw at 3.5, 6, 11 and 12 months of age.
  rMenB + OMV NZ vaccine: 3 doses (2.5, 3.5, 5 months if age) plus booster (11 months of age)
- B_3h5_11b: Subjects, approximately 3.5 months of age, received 2 dose primary vaccination of rMenB+OMV NZ at 3.5 and 5 months of age, followed by a booster dose at 11 months of age. Blood draw at 5, 11 and 12 months of age.
  rMenB + OMV NZ vaccine: 2 doses (3.5, 5 months of age) plus booster (11 months of age)
- B_68_11b: Subjects, approximately 6 months of age, received 2 dose primary vaccination of rMenB+OMV NZ at 6 and 8 months of age, followed by a booster dose at 11 months of age. Blood draw at 8, 9, 11 and 12 months of age.
  rMenB + OMV NZ vaccine: 2 doses (6, 8 months of age) plus booster (11 months of age)
Arm/Group | B_2h3h5_11b | B_3h5_11b | B_68_11b
Number analyzed (Participants) | 119 | 115 | 118
Titers
  H44/76 1 month after 1st vacc; N=117,115,117 | 4.19 [3.29 to 5.35] | 5.7 [4.41 to 7.37] | 9.83 [7.59 to 13]
  5/99 1 month after 1st vacc | 20 [15 to 27] | 30 [22 to 42] | 37 [27 to 52]
  NZ98/254 1 month after 1st vacc; N=118,114,117 | 2.87 [2.32 to 3.54] | 2.48 [1.98 to 3.11] | 2.84 [2.28 to 3.55]
  M10713 1 month after 1st vacc; N=95,99,95 | 2.59 [1.86 to 3.6] | 1.69 [1.21 to 2.36] | 1.62 [1.15 to 2.28]

7. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 4 or hSBA Titers ≥ 5 and hSBA ≥ 8 After First Infant Vaccination With rMenB+OMV
Description: Immunogenicity was assessed in terms of percentages of subjects with hSBA titers ≥ 4 against N meningitidis serogroup B strains H44/76, 5/99, NZ98/254, hSBA titers ≥ 5 against strain M10713 and hSBA titers ≥ 8 against strains H44/76, 5/99, NZ98/254, M10713 after the first infant vaccination in groups B_2h3h5_11b, B_3h5_11b and B_68_11b (at 3.5, 5, and 8 months of age respectively). Analysis was done on FAS-post first dose.
Time Frame: Post- first dose (1 month for B_2h3h5_11b, 1.5 month for B_3h5_11b and 2 months for B_68_11b after 1st vaccination)
Population: FAS-post first dose
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- B_3h5_11b: Subjects, approximately 3.5 months of age, received 2 dose primary vaccination of rMenB+OMV NZ at 3.5 and 5 months of age, followed by a booster dose at 11 months of age. Blood draw at 5, 11 and 12 months of age.
  rMenB + OMV NZ vaccine: 2 doses (3-1/2, 5 months of age) plus booster (11 months of age)
Arm/Group | B_2h3h5_11b | B_3h5_11b | B_68_11b
Number analyzed (Participants) | 119 | 115 | 118
Percentages of subjects
  H44/76 (hSBA≥ 4; Post 1st vacc; N=117,115,117) | 62 [52 to 70] | 72 [63 to 80] | 82 [74 to 89]
  5/99 (hSBA≥ 4; Post 1st vacc) | 91 [84 to 95] | 95 [89 to 98] | 92 [86 to 96]
  NZ98/254 (hSBA≥ 4; Post 1st vacc; N=118,114,117) | 43 [34 to 53] | 39 [30 to 48] | 41 [32 to 50]
  M10713 (hSBA≥ 5; Post1st vacc; N=95,99,95) | 31 [21 to 41] | 18 [11 to 27] | 17 [10 to 26]
  H44/76 (hSBA≥ 8; Post 1st vacc; N=117,115,117) | 25 [17 to 34] | 38 [29 to 48] | 58 [49 to 67]
  5/99 (hSBA≥ 8; Post1st vacc) | 82 [73 to 88] | 90 [82 to 94] | 86 [79 to 92]
  NZ98/254 (hSBA≥ 8; 1st vacc; N=118,114,117) | 13 [7 to 20] | 7 [3 to 13] | 13 [7 to 20]
  M10713 (hSBA≥ 8; Post1st vacc; N=95,99,95) | 21 [13 to 31] | 15 [9 to 24] | 13 [7 to 21]

8. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 4 or hSBA Titers ≥ 5 and hSBA ≥ 8 Following a Booster Dose of rMenB+OMV Vaccination
Description: Immunogenicity was assessed in terms of percentages of subjects with hSBA titers ≥ 4 against N meningitidis serogroup B strains H44/76, 5/99, NZ98/254; hSBA titers ≥ 5 against strain M10713; hSBA titers ≥ 8 against strains H44/76, 5/99, NZ98/254, M10713; following a booster dose of rMenB+OMV NZ given at 11 months of age (4th dose for B_2h3h5_11 and 3rd dose for B_3h5_11 and B_68_11). Analysis was done on FAS-booster.
Time Frame: 1 month post-booster dose
Population: FAS-booster
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- B_3h5_11: Subjects, approximately 3.5 months of age, received 2 dose primary vaccination of rMenB+OMV NZ at 3.5 and 5 months of age, followed by a booster dose at 11 months of age.
  rMenB + OMV NZ vaccine: 2 doses (3-1/2, 5 months of age) plus booster (11 months of age)
Arm/Group | B_2h3h5_11 | B_3h5_11 | B_68_11
Number analyzed (Participants) | 233 | 228 | 239
Percentages of subjects
  H44/76 (hSBA≥ 4, after booster; N=233,227,238) | 100 [98 to 100] | 100 [98 to 100] | 100 [98 to 100]
  5/99 (hSBA≥ 4, after booster) | 100 [98 to 100] | 100 [98 to 100] | 100 [98 to 100]
  NZ98/254 (hSBA≥ 4, after booster; N=231,226,236) | 100 [98 to 100] | 99 [96 to 100] | 100 [98 to 100]
  M10713 (hSBA≥ 5, after booster; N=203,181,193) | 83 [77 to 88] | 87 [81 to 91] | 83 [77 to 88]
  H44/76 (hSBA≥ 8, after booster; N=233,227,238) | 100 [98 to 100] | 100 [98 to 100] | 100 [98 to 100]
  5/99 (hSBA≥ 8, after booster) | 100 [98 to 100] | 100 [98 to 100] | 100 [98 to 100]
  NZ98/254 (hSBA≥ 8, after booster; N=231,226,236) | 95 [91 to 97] | 95 [91 to 98] | 97 [95 to 99]
  M10713 (hSBA≥ 8, after booster; N=203,181,193) | 78 [72 to 84] | 83 [77 to 89] | 74 [67 to 80]

9. Secondary Outcome: Antibody Persistence in Terms of Percentages of Subjects With hSBA Titers ≥ 4 or hSBA Titers ≥ 5 (M10713) and hSBA ≥ 8 Following 2 or 3-dose Primary Series of Vaccination With rMenB+OMV NZ
Description: Persistence of bactericidal antibodies at 11 months of age was assessed in terms of percentages of subjects with hSBA titers ≥ 4 against N meningitidis serogroup B strains H44/76, 5/99, NZ98/254; hSBA titers ≥ 5 against strain M10713; hSBA titers ≥ 8 against strains H44/76, 5/99, NZ98/254, M10713 in subjects who previously received a primary series of 2 or 3-doses of rMenB+OMV NZ vaccine. Analysis was done on FAS-persistence.
Time Frame: 11 months of age (persistence)
Population: FAS-persistence
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | B_2h3h5_11 | B_3h5_11 | B_68_11
Number analyzed (Participants) | 235 | 233 | 238
Percentages of subjects
  H44/76 (hSBA≥ 4; 11 months of age; N=235,232,237) | 87 [82 to 91] | 86 [81 to 90] | 100 [98 to 100]
  5/99 (hSBA≥ 4; 11 months of age; N=234,230,235) | 100 [98 to 100] | 93 [89 to 96] | 100 [98 to 100]
  NZ98/254 hSBA≥ 4; 11 months of age; N=233,233,238) | 54 [47 to 60] | 41 [34 to 47] | 90 [85 to 93]
  M10713 (hSBA≥ 5; 11 months of age; N=199,177,188) | 33 [26 to 40] | 23 [17 to 30] | 42 [35 to 49]
  H44/76 (hSBA≥ 8; 11 months of age; N=235,232,237) | 64 [58 to 70] | 60 [53 to 66] | 96 [93 to 98]
  5/99 (hSBA≥ 8; 11 months of age; N=234,230,235) | 94 [91 to 97] | 87 [82 to 91] | 99 [97 to 100]
  NZ98/254 hSBA≥ 8; 11 months of age; N=233,233,238) | 36 [30 to 43] | 12 [8 to 17] | 65 [58 to 71]
  M10713 (hSBA≥ 8; 11 months of age; N=199,177,188) | 24 [18 to 30] | 16 [11 to 22] | 36 [29 to 43]

10. Secondary Outcome: Antibody Persistence in Terms of Geometric Mean Titers Following 2 or 3-dose Primary Series of Vaccination With rMenB+OMV NZ
Description: Persistence of bactericidal antibodies at 11 months of age was assessed in terms of GMTs against N meningitidis serogroup B indicator strains in subjects who previously received a primary series of 2 or 3-doses of rMenB+OMV NZ. Analysis was done on FAS-persistence.
Time Frame: 11 months of age (persistence)
Population: FAS-persistence
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | B_2h3h5_11 | B_3h5_11 | B_68_11
Number analyzed (Participants) | 235 | 233 | 238
Titers
  H44/76 (Baseline; N=111,113,120) | 1.31 [1.09 to 1.57] | 1.34 [1.11 to 1.62] | 1.58 [1.32 to 1.9]
  H44/76 (11 moa; N=235,232,237)) | 12 [9.64 to 14] | 12 [9.39 to 14] | 67 [55 to 82]
  5/99 (Baseline; N=113,112,120) | 1.15 [1.02 to 1.3] | 1.16 [1.02 to 1.32] | 0.97 [0.85 to 1.09]
  5/99 (11 moa; N=234,230,235) | 98 [78 to 124] | 50 [39 to 63] | 285 [225 to 363]
  NZ98/254 (Baseline; N=113,113,122) | 1.07 [0.99 to 1.15] | 1.04 [0.96 to 1.12] | 1 [0.93 to 1.07]
  NZ98/254 (11 moa; N=233,233,238) | 4.57 [3.66 to 5.71] | 2.68 [2.13 to 3.38] | 12 [9.79 to 15]
  M10713 (Baseline; N=84,64,88) | 2.36 [1.75 to 3.2] | 1.52 [1.07 to 2.17] | 1.29 [0.95 to 1.76]
  M10713 (11 moa; N=199,177,188) | 2.55 [1.89 to 3.43] | 1.98 [1.45 to 2.71] | 3.62 [2.66 to 4.94]

11. Secondary Outcome: Geometric Mean ELISA Concentrations Against Vaccine Antigen 287-953 Following 2 or 3-dose Primary Series and Booster Dose of Vaccination With rMenB+OMV NZ
Description: Immunogenicity was assessed in terms of Geometric mean ELISA concentrations (GMCs) against N meningitidis serogroup B vaccine antigen 287-953, following 2 or 3 dose primary series and booster dose of rMenB+OMV NZ. Analysis was done on FAS-persistence and FAS-booster.
Time Frame: 1 month after primary vaccination, pre-booster vaccination (persistence) and 1 month after booster vaccination
Population: FAS-persistence and FAS-booster
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | B_2h3h5_11 | B_3h5_11 | B_68_11
Number analyzed (Participants) | 218 | 225 | 221
IU/mL
  1 month after primary vaccination (N=212,215,212) | 4688 [3884 to 5660] | 3152 [2594 to 3831] | 4682 [3850 to 5694]
  Pre-booster vaccination (N=213,220,215) | 474 [395 to 569] | 291 [241 to 351] | 1270 [1052 to 1533]
  1 month after booster dose | 5900 [5047 to 6898] | 6062 [5150 to 7135] | 5898 [5016 to 6934]

12. Secondary Outcome: Geometric Mean ELISA Concentrations Against Vaccine Antigen 287-953 After a Two Dose Catch-up rMenB+OMV NZ Immunization Series in Children 2-10 Years of Age
Description: Immunogenicity was assessed in terms of Geometric mean ELISA concentrations (GMCs) against N meningitidis serogroup B vaccine antigen 287-953, after a two dose catch-up immunization series with rMenB+OMV NZ in children 2-10 years of age. Analysis was done on FAS-primary series.
Time Frame: 1 month after second vaccination
Population: FAS-primary series
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | B_02
Number analyzed (Participants) | 389
IU/mL | 2333 [2124 to 2562]

13. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 8 Against Serogroup C Following Concomitant Administration of rMenB+OMV NZ With MenC-CRM or MenC-CRM Alone
Description: Non-inferiority of MenC-CRM was determined following co-administration of MenC-CRM and rMenB+OMV NZ or MenC-CRM alone at 3 and 5 months and booster dose at 12 months, as measured by the percentages of subjects achieving hSBA titers ≥ 8 against serogroup C. Analysis was done on PPS-primary series and PPS-booster.
Time Frame: Baseline, 1 month after second vaccination and 1 month after booster vaccination
Population: PPS-primary series and PPS-booster.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | BC_35_12 | C_35_12
Number analyzed (Participants) | 85 | 72
Percentages of subjects
  Serogroup C (1 month after 2nd vacc) | 99 [94 to 100] | 100 [95 to 100]
  Serogroup C (1 month after booster vacc; N=70,47) | 100 [95 to 100] | 100 [92 to 100]
Statistical Analysis 1: Comparison: BC_35_12 vs C_35_12; Non-inferiority of MenC-CRM was determined following co-administration of MenC-CRM and rMenB+OMV NZ vs MenC-CRM control group at 1 month after 2nd vaccination for serogroup C; Test type: Non-Inferiority or Equivalence — Non-inferiority; Miettinen and Nurminen method; Vaccine group difference = -1, 95% CI 2-sided [-6.4 to 3.9]
Statistical Analysis 2: Comparison: BC_35_12 vs C_35_12; Non-inferiority of MenC-CRM was determined following co-administration of MenC-CRM and rMenB+OMV NZ vs MenC-CRM control group at 1 month after booster vaccination for serogroup C; Test type: Non-Inferiority or Equivalence — Non-inferiority; Miettinen and Nurminen method; Vaccine group difference = 0, 95% CI 2-sided [-5.2 to 7.6]

14. Secondary Outcome: GMTs Following Concomitant Administration of rMenB+OMV NZ With MenC-CRM or MenC-CRM Alone
Description: Immunogenicity was assessed in terms of GMTs against N meningitidis serogroup C strain following co-administration of MenC-CRM and rMenB+OMV NZ or MenC-CRM alone at 3 and 5 months and booster dose at 12 months. Analysis was done on FAS-primary series and FAS-booster.
Time Frame: 1 month after second vaccination, 1 month after booster vaccination
Population: FAS-primary series and FAS-booster
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | BC_35_12 | C_35_12
Number analyzed (Participants) | 102 | 88
Titers
  1 month after 2nd vacc | 568 [461 to 701] | 905 [718 to 1141]
  Pre-booster vacc (N=92,75) | 36 [28 to 47] | 56 [41 to 77]
  1 month after booster vacc (N=99,92) | 1201 [991 to 1456] | 1724 [1350 to 2201]

15. Secondary Outcome: GMTs Following Concomitant Administration of rMenB+OMV NZ With MenC-CRM or MenC-CRM Alone - Persistence
Description: Immunogenicity was assessed in terms of GMTs against N meningitidis serogroup C strain following co-administration of MenC-CRM and rMenB+OMV NZ or MenC-CRM alone at 3 and 5 months and booster dose at 12 months. Analysis was done on FAS-persistence.
Time Frame: Pre-booster vaccination (persistence; 12 months of age)
Population: FAS-persistence
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- BC_35_12: Subjects, 3 months of age received rMenB+OMV NZ + MenC-CRM and Synflorix concomitantly at 3, 5 and 12 months of age and an additional dose of Synflorix alone dose at 7 months of age.
  Meningococcal C oligosaccharide conjugated vaccine: Schedule 3, 5, 7 12, Meningococcal C oligosaccharide conjugated vaccine
  Pneumococcal polysaccharide conjugate vaccine, 10 valent adsorbed.: Schedule 3, 5, 7, 12 Pneumococcal polysaccharide conjugate vaccine, 10 valent adsorbed.
  rMenB + OMV NZ vaccine: Schedule 3, 5 12 rMenB + OMV vaccine
- C_35_12: Subjects, 3 months of age received MenC-CRM and Synflorix concomitantly at 3, 5 and 12 months of age and an additional dose of Synflorix alone at 7 months of age and rMenB+OMV NZ alone at 13 ad 15 months of age.
  Meningococcal C oligosaccharide conjugated vaccine: Schedule 3, 5, 7 12, Meningococcal C oligosaccharide conjugated vaccine
  Pneumococcal polysaccharide conjugate vaccine, 10 valent adsorbed.: Schedule 3, 5, 7, 12 Pneumococcal polysaccharide conjugate vaccine, 10 valent adsorbed.
  rMenB + OMV NZ vaccine: Schedule 13,15 rMenB + OMV vaccine
Arm/Group | BC_35_12 | C_35_12
Number analyzed (Participants) | 108 | 93
Titers | 36 [28 to 46] | 56 [41 to 75]

16. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 4 or hSBA Titers ≥ 5 (M10713) and hSBA ≥ 8 Following Concomitant Administration of rMenB+OMV NZ With MenC-CRM
Description: Immunogenicity was assessed in terms of percentages of subjects with hSBA titers ≥ 4 against N meningitidis serogroup B strains H44/76, 5/99, NZ98/254; hSBA titers ≥ 5 against strain M10713; hSBA titers ≥ 8 against strains H44/76, 5/99, NZ98/254, M10713; following co-administration of MenC-CRM and rMenB+OMV NZ at 3 and 5 months and a booster at 12 months. Analysis was done on FAS-primary series and FAS-booster.
Time Frame: 1 month after second vaccination and 1 month after booster vaccination
Population: FAS-primary series and FAS-booster
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | BC_35_12
Number analyzed (Participants) | 119
Percentages of subjects
  H44/76 (hSBA≥4; 1 month after 2nd vacc) | 97 [92 to 99]
  H44/76 (hSBA≥4; 1 month after booster vacc; N=114) | 100 [97 to 100]
  5/99 (hSBA≥4; 1 month after 2nd vacc) | 96 [90 to 99]
  5/99 (hSBA≥4; 1 month after booster vacc; N=113) | 97 [92 to 99]
  NZ98/254 (hSBA≥4; 1 month after 2nd vacc; N=118) | 95 [89 to 98]
  NZ98/254 (hSBA≥4; 1 mo after booster vacc; N=114) | 97 [93 to 99]
  M10713 (hSBA≥5; 1 month after 2nd vacc; N=98) | 68 [58 to 77]
  M10713 (hSBA≥5; 1 month after booster vacc; N=101) | 67 [57 to 76]
  H44/76 (hSBA≥8; 1 month after 2nd vacc) | 97 [92 to 99]
  H44/76 (hSBA≥8; 1 month after booster vacc; N=114) | 99 [95 to 100]
  5/99 (hSBA≥8; 1 month after 2nd vacc) | 96 [90 to 99]
  5/99 (hSBA≥8; 1 month after booster vacc; N=113) | 97 [92 to 99]
  NZ98/254 (hSBA≥8; 1 month after 2nd vacc; N=118) | 87 [80 to 93]
  NZ98/254 (hSBA≥8; 1 mo after booster vacc; N=114) | 95 [89 to 98]
  M10713 (hSBA≥8; 1 month after 2nd vacc; N=98) | 60 [50 to 70]
  M10713 (hSBA≥8; 1 month after booster vacc; N=101) | 61 [51 to 71]

17. Secondary Outcome: GMTs Against N. Meningitidis Serogroup B Strains Following Concomitant Administration of rMenB+OMV NZ With MenC-CRM
Description: Immunogenicity was assessed in terms of GMTs against N meningitidis serogroup C strain following co-administration of MenC-CRM and rMenB+OMV NZ at 3 and 5 months and booster dose at 12 months. Analysis was done on FAS-persistence and FAS-booster.
Time Frame: 1 month after second vaccination, pre-booster vaccination and 1 month after booster vaccination
Population: FAS-persistence and FAS-booster
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | BC_35_12
Number analyzed (Participants) | 115
Titers
  H44/76 (1 month after 2nd vacc) | 226 [179 to 284]
  H44/76 (Pre-booster vacc) | 16 [13 to 20]
  H44/76 (1 month after booster vacc; N=114) | 239 [198 to 288]
  5/99 (1 month after 2nd vacc) | 555 [409 to 753]
  5/99 (Pre-booster vacc) | 55 [42 to 72]
  5/99 (1 month after booster vacc; N=113) | 1623 [1210 to 2176]
  NZ98/254 (1 month after 2nd vacc; N=114) | 27 [21 to 34]
  NZ98/254 (Pre-booster vacc; N=115) | 2.63 [2.21 to 3.14]
  NZ98/254 (1 month after booster vacc; N=114) | 68 [54 to 86]
  M10713 (1 month after 2nd vacc; N=89) | 9.81 [7.06 to 14]
  M10713 (Pre-booster vacc; N=110) | 2.2 [1.72 to 2.82]
  M10713 (1 month after booster vacc; N=101) | 11 [7.72 to 15]

18. Secondary Outcome: Geometric Mean ELISA Concentrations Against Vaccine Antigen 287-953 Following Concomitant Administration of rMenB+OMV NZ With MenC-CRM
Description: Immunogenicity was assessed in terms of Geometric mean ELISA concentrations against N meningitidis serogroup B vaccine antigen 287-953, following co-administration of MenC-CRM and rMenB+OMV NZ at 3 and 5 months and booster dose at 12 months. Analysis was done on FAS-primary and FAS-booster.
Time Frame: 1 month after second vaccination, pre-booster vaccination and 1 month after booster vaccination
Population: FAS-primary and FAS-booster
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BC_35_12
Number analyzed (Participants) | 116
IU/mL
  1 month after 2nd vacc | 2125 [1595 to 2830]
  Pre-booster vacc (N=111) | 194 [164 to 230]
  1 month after booster vacc (N=113) | 4281 [3411 to 5372]

19. Secondary Outcome: Geometric Mean ELISA Concentrations Against Vaccine Antigen 287-953 Following Concomitant Administration of rMenB+OMV NZ With MenC-CRM - Persistence
Description: Immunogenicity was assessed in terms of GMTs against Geometric mean ELISA concentrations against N meningitidis serogroup B vaccine antigen 287-953, following co-administration of MenC-CRM and rMenB+OMV NZ at 3 and 5 months and booster dose at 12 months. Analysis was done on FAS-persistence.
Time Frame: Pre-booster vaccination (persistence; 12 months of age)
Population: FAS-persistence
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BC_35_12
Number analyzed (Participants) | 115
IU/mL | 196 [166 to 231]

20. Secondary Outcome: Number of Subjects Who Reported Immediate Reactions Within 30 Minutes After Any Vaccination With rMenB+OMV NZ
Description: Safety was assessed in terms of number of subjects who reported immediate reactions within 30 minutes following a 4-dose regimen (2.5, 3.5, 5 and 11 months) or a 3-dose regimen (3.5, 5 and 11 months or 6, 8 and 11 months) of rMenB+OMV NZ. Analysis was done on solicited safety set.
Time Frame: Within 30 minutes after any vaccination
Population: Solicited safety set.
Measure: Number; unit: Number of subjects
Arm/Group | B_2h3h5_11b | B_3h5_11b | B_68_11b
Number analyzed (Participants) | 252 | 249 | 250
Number of subjects
  Tenderness | 13 | 9 | 9
  Erythema | 19 | 19 | 7
  Induration | 4 | 3 | 2
  Swelling | 1 | 2 | 1
  Change in eating habits | 0 | 2 | 1
  Sleepiness | 1 | 2 | 3
  Unusual crying | 4 | 3 | 4
  Vomiting | 1 | 0 | 0
  Diarrhea | 0 | 0 | 1
  Irritability | 1 | 2 | 1
  Rash | 0 | 1 | 1
  Fever (≥38°C) | 3 | 2 | 2
  Medic. used for pain (N=252,248,250) | 0 | 0 | 0
  Medically-attended fever | 0 | 0 | 0
  Medic. used to treat high temp. (N=252,248,250) | 1 | 1 | 0
  Medic. used to prevent high temp. (N=252,248,250) | 0 | 0 | 0

21. Secondary Outcome: Number of Subjects With Solicited Local and Systemic Adverse Events (AEs) Following a 3 or 4-dose Regimen of rMenB+OMV NZ
Description: Safety was assessed in terms of number of subjects with solicited local and systemic AEs after any vaccination following a 4-dose regimen (2.5, 3.5, 5 and 11 months) or as a 3-dose regimen (3.5, 5 and 11 months or 6, 8 and 11 months) of rMenB+OMV NZ. Analysis was done on solicited safety set.
Time Frame: Day 1 to day 7 after any vaccination
Population: Solicited safety set
Measure: Number; unit: Number of subjects
Arm/Group | B_2h3h5_11 | B_3h5_11 | B_68_11
Number analyzed (Participants) | 247 | 243 | 246
Number of subjects
  Any local (N=245,241,244) | 226 | 213 | 202
  Tenderness (N=245,241,244) | 200 | 174 | 166
  Erythema (N=245,241,244) | 164 | 156 | 157
  Induration (N=245,241,244) | 161 | 117 | 121
  Swelling (N=245,241,244) | 120 | 75 | 84
  Any systemic (N=245,241,244) | 238 | 236 | 233
  Change in eating habits (N=245,241,244) | 141 | 112 | 121
  Sleepiness (N=245,241,244) | 186 | 152 | 143
  Irritability (N=245,241,244) | 180 | 156 | 151
  Vomiting (N=245,241,244) | 65 | 39 | 55
  Diarrhea (N=245,241,244) | 91 | 69 | 74
  Rash (N=245,241,244) | 23 | 21 | 22
  Unusual Crying (N=245,241,244) | 198 | 186 | 156
  Fever (≥38°C) (N=245,241,244) | 197 | 189 | 184
  Medic. used for pain (N=245,241,244) | 129 | 110 | 109
  Medic. used to prevent high temp. (N=245,241,244) | 97 | 94 | 99
  Medic. used to treat high temp. (N=245,242,244) | 193 | 186 | 177
  Medically-attended fever | 16 | 10 | 15

22. Secondary Outcome: Number of Subjects Who Reported Immediate Reactions Within 30 Minutes After Any Vaccination - Groups B_02_2_5 and B_02_6_10
Description: Safety was assessed in terms of number of subjects with solicited local and systemic AEs after any vaccination in subjects aged 2 - 10 years who received 2 catch-up doses of rMenB+OMV NZ, each at 0 and 2 months. Analysis was done on solicited safety set.
Time Frame: Within 30 minutes after any vaccination
Population: Solicited safety set
Measure: Number; unit: Number of subjects
Arm/Group | B_02_2_5 | B_02_6_10
Number analyzed (Participants) | 104 | 300
Number of subjects
  Pain | 6 | 17
  Erythema | 6 | 2
  Induration | 1 | 3
  Swelling | 2 | 2
  Chills (N=0,300) | NA — Solicited AE not applicable for this age-group. | 2
  Change in eating habits (N=104,0) | 0 | NA — Solicited AE not applicable for this age-group.
  Sleepiness (N=104,0) | 0 | NA — Solicited AE not applicable for this age-group.
  Irritability (N=104,0) | 1 | NA — Solicited AE not applicable for this age-group.
  Vomiting (N=104,0) | 0 | NA — Solicited AE not applicable for this age-group.
  Nausea (N=0,300) | NA — Solicited AE not applicable for this age-group. | 2
  Malaise (N=0,300) | NA — Solicited AE not applicable for this age-group. | 4
  Diarrhoea (N=104,0) | 0 | NA — Solicited AE not applicable for this age-group.
  Headache | 0 | 1
  Rash | 0 | 0
  Arthralgia | 0 | 1
  Myalgia (N=0,300) | NA — Solicited AE not applicable for this age-group. | 5
  Fever (≥38°C) | 0 | 0
  Medic. used for pain | 0 | 1
  Medic. used to prevent high temp. | 0 | 1
  Medic. used to treat high temp | 0 | 0
  Medically-attended fever | 0 | 0

23. Secondary Outcome: Number of Subjects With Solicited Local and Systemic AEs in Groups B_02_2_5 and B_02_6_10
Description: Safety was assessed in terms of number of subjects with solicited local and systemic AEs after any vaccination in subjects aged 2- 10 years who received 2 catch-up doses of rMenB+OMV NZ, each at 0 and 2 months. Analysis was done on solicited safety set.
Time Frame: Day 1 to day 7 after any vaccination
Population: Solicited safety set
Measure: Number; unit: Number of subjects
Arm/Group | B_02_2_5 | B_02_6_10
Number analyzed (Participants) | 102 | 299
Number of subjects
  Any Local (N=100,297) | 99 | 287
  Pain (N=100,297) | 98 | 287
  Erythema (N=100,297) | 58 | 179
  Induration (N=100,297) | 41 | 123
  Swelling (N=100,297) | 50 | 146
  Any systemic (N=100,297) | 78 | 205
  Chills (N=0,296) | NA — Solicited AE not applicable for this age-group. | 45
  Change in eating habits (N=100,0) | 35 | NA — Solicited AE not applicable for this age-group.
  Sleepiness (N=100,0) | 39 | NA — Solicited AE not applicable for this age-group.
  Irritability (N=100,0) | 49 | NA — Solicited AE not applicable for this age-group.
  Malaise (N=0,296) | NA — Solicited AE not applicable for this age-group. | 114
  Vomiting (N=100,0) | 7 | NA — Solicited AE not applicable for this age-group.
  Nausea (N=0,296) | NA — Solicited AE not applicable for this age-group. | 36
  Diarrhea (N=100,0) | 12 | NA — Solicited AE not applicable for this age-group.
  Headache (N=100,296) | 7 | 89
  Rash (N=100,296) | 9 | 20
  Arthralgia (N=100,296) | 35 | 49
  Myalgia (N=0,296) | NA — Solicited AE not applicable for this age-group. | 126
  Fever (≥38°C) (N=100,296) | 20 | 41
  Medic. used for pain (N=100,296) | 48 | 158
  Medic. used to prevent high temp. (N=100,296) | 7 | 44
  Medic. used to treat high temp. (N=100,296) | 20 | 54
  Medically-attended fever | 0 | 7

24. Secondary Outcome: Number of Subjects Who Reported Immediate Reactions Within 30 Minutes After Any rMenB+OMV NZ or MenC-CRM Vaccination
Description: Safety was assessed in terms of number of subjects with solicited local and systemic AEs after any vaccination with rMenB+OMV NZ or MenC-CRM. Analysis was done on solicited safety set.
Time Frame: Within 30 minutes after any vaccination
Population: Solicited safety set
Measure: Number; unit: Number of subjects
Arm/Group | BC_35_12 | C_35_12
Number analyzed (Participants) | 126 | 124
Number of subjects
  Tenderness (rMenB+OMV NZ) (N=126,0) | 7 | NA — Subjects in this group did not receive rMenB+OMV NZ vaccination.
  Erythema (rMenB+OMV NZ) (N=126,0) | 3 | NA — Subjects in this group did not receive rMenB+OMV NZ vaccination.
  Induration (rMenB+OMV NZ) (N=126,0) | 1 | NA — Subjects in this group did not receive rMenB+OMV NZ vaccination.
  Swelling (rMenB+OMV NZ) (N=126,0) | 0 | NA — Subjects in this group did not receive rMenB+OMV NZ vaccination.
  Tenderness (MenC-CRM) | 5 | 5
  Erythema (MenC-CRM) | 4 | 5
  Induration (MenC-CRM) | 0 | 0
  Swelling (MenC-CRM) | 0 | 0
  Change in eating habits | 0 | 0
  Sleepiness | 0 | 0
  Unusual crying | 0 | 0
  Irritability | 0 | 0
  Vomiting | 1 | 0
  Diarrhea | 0 | 0
  Rash | 0 | 0
  Fever (≥38°C) | 1 | 0
  Medic. used for pain | 0 | 0
  Medic. used to prevent high temp. | 0 | 0
  Medic. used to treat high temp. | 0 | 0
  Medically-attended fever | 0 | 0

25. Secondary Outcome: Number of Subjects With Solicited Local and Systemic AEs in Groups BC_35_12 and C_35_12 After Any rMenB+OMV NZ or MenC-CRM Vaccination
Description: as for outcome 24
Time Frame: Day 1 to day 7 after any vaccination
Population: Solicited safety set
Measure: Number; unit: Number of subjects
Arm/Group | BC_35_12 | C_35_12
Number analyzed (Participants) | 124 | 117
Number of subjects
  Any local rMenB + OMZ NV | 107 | NA — Subjects in this group did not receive rMenB+OMV NZ vaccination.
  Any local MenC-CRM | 104 | 79
  Any systemic | 123 | 106
  Tenderness (rMenB+OMV NZ) (N=123,0) | 105 | NA — Subjects in this group did not receive rMenB+OMV NZ vaccination.
  Erythema (rMenB+OMV NZ) (N=123,0) | 48 | NA — Subjects in this group did not receive rMenB+OMV NZ vaccination.
  Induration (rMenB+OMV NZ) (N=123,0) | 37 | NA — Subjects in this group did not receive rMenB+OMV NZ vaccination.
  Swelling (rMenB+OMV NZ) (N=123,0) | 21 | NA — Subjects in this group did not receive rMenB+OMV NZ vaccination.
  Tenderness (MenC-CRM) (N=123,117) | 104 | 74
  Erythema (MenC-CRM) (N=123,117) | 25 | 24
  Induration (MenC-CRM) (N=123,117) | 10 | 26
  Swelling (MenC-CRM) (N=123,117) | 12 | 21
  Change in eating habits (N=123,117) | 67 | 47
  Sleepiness (N=123,117) | 93 | 78
  Unusual crying (N=123,117) | 105 | 87
  Irritability (N=123,117) | 95 | 66
  Vomiting (N=123,117) | 29 | 27
  Diarrhea (N=123,117) | 41 | 40
  Rash (N=123,117) | 8 | 4
  Fever (≥38°C) (N=123,117) | 97 | 45
  Medic. used for pain (N=123,117) | 102 | 69
  Medic. used to prevent high temp. | 49 | 25
  Medic. used to treat high temp. | 90 | 40
  Medically-attended fever | 7 | 12

26. Secondary Outcome: Number of Subjects Reporting Unsolicited AEs Following Any Vaccination With rMenB+OMV NZ in Groups B_2h3h5_11, B_3h5_11 and B_68_11
Description: Safety was assessed in terms of number of subjects reporting any unsolicited AEs (day 1-7 after any vaccination), serious adverse events (SAEs), medically attended AEs, AEs leading to premature withdrawal from the study (collected throughout the study period) following any vaccination with rMenB+OMV. Analysis was done on unsolicited safety set.
Time Frame: Until 12 months of age; Day 1 to day 7 (All AEs)
Population: Unsolicited safety set
Measure: Number; unit: Number of subjects
Arm/Group | B_2h3h5_11b | B_3h5_11b | B_68_11b
Number analyzed (Participants) | 252 | 249 | 250
Number of subjects
  All AEs (days 1-7) | 200 | 186 | 196
  At least possible related AEs | 88 | 41 | 62
  SAEs | 15 | 18 | 9
  At least possibly related SAEs | 1 | 1 | 1
  Medically attended AEs | 178 | 179 | 182
  AEs leading to premature withdrawal | 1 | 1 | 0
  Deaths | 0 | 0 | 0

27. Secondary Outcome: Number of Subjects Reporting Unsolicited AEs Following Any Vaccination With rMenB+OMV NZ in Groups B_02_2_5 and B_02_6_10
Description: Safety was assessed in terms of number of subjects reporting any unsolicited AEs (day 1-7 after any vaccination), serious adverse events (SAEs), medically attended AEs, AEs leading to premature withdrawal from the study (collected throughout the study period) following any vaccination with rMenB+OMV NZ. Analysis was done on unsolicited safety set.
Time Frame: Day 1 to day 7 (All AEs). Throughout the study period (SAEs, medically attended or leading to premature withdrawal AEs)
Population: Unsolicited safety set
Measure: Number; unit: Number of subjects
Arm/Group | B_02_2_5 | B_02_6_10
Number analyzed (Participants) | 104 | 300
Number of subjects
  All AEs (days 1-7) | 58 | 101
  At least possible related AEs | 16 | 24
  SAEs | 1 | 2
  At least possibly related SAEs | 0 | 0
  Medically attended AEs | 42 | 74
  AEs leading to premature withdrawal | 0 | 0
  Deaths | 0 | 0

28. Secondary Outcome: Number of Subjects Reporting Unsolicited AEs Following Any Vaccination With rMenB+OMV NZ in Group BC_35_12 and C_35_12
Description: Safety was assessed in terms of number of subjects reporting any unsolicited AEs (day 1-7 after any vaccination), serious adverse events (SAEs), medically attended AEs, AEs leading to premature withdrawal from the study (collected throughout the study period) following any vaccination with rMenB+OMV NZ or MenC-CRM. Analysis was done on unsolicited safety set.
Time Frame: Day 1 to Day 301 for BC_35_12 and C_35_12, Day 302 to Day 391 for C_35_12; Day 1 to day 7 (All AEs)
Population: Unsolicited safety set
Measure: Number; unit: Number of subjects
Arm/Group | BC_35_12 | C_35_12
Number analyzed (Participants) | 126 | 123
Number of subjects
  All AEs (days 1-7) | 103 | 90
  At least possibly related AEs | 14 | 12
  SAEs | 5 | 7
  At least possibly related SAEs | 0 | 0
  Medically attended AEs | 99 | 85
  AEs leading to premature withdrawal | 0 | 0
  Deaths | 0 | 0

ADVERSE EVENTS:
Time Frame: Till 12 months of age for groups B_2h3h5_11, B_3h5_11 and B_68_11; Day 1 to Day 91 for groups B02_2_5 and B02_6_10; Day 1 to Day 301 for group BC_35_12; Day 1 to Day 391 for group C_35_12.
Description: All solicited AEs were collected by systematic assessment and unsolicited AEs were collected by non-systematic assessment.
Groups:
- TOTAL: All subjects in the safety population.
Arm/Group | B_2h3h5_11 | B_3h5_11 | B_68_11 | B_02_2_5 | B_02_6_10 | BC_35_12 | C_35_12 | TOTAL
Serious Adverse Events (participants affected / at risk) | 15/252 | 18/249 | 9/250 | 1/104 | 2/300 | 5/126 | 8/123 | 58/1404
Other Adverse Events (participants affected / at risk) | 246/252 | 240/249 | 245/250 | 100/104 | 288/300 | 124/126 | 115/123 | 1358/1404
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B_2h3h5_11 (N=252) | B_3h5_11 (N=249) | B_68_11 (N=250) | B_02_2_5 (N=104) | B_02_6_10 (N=300) | BC_35_12 (N=126) | C_35_12 (N=123) | TOTAL (N=1404)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
CONGENITAL CENTRAL NERVOUS SYSTEM ANOMALY (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
GLAUCOMA (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
ALLERGIC COLITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
FOOD POISONING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
PYREXIA (General disorders) | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 5
ATYPICAL PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
BRONCHIOLITIS (Infections and infestations) | 1 | 2 | 3 | 0 | 0 | 2 | 1 | 9
BRONCHITIS (Infections and infestations) | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 5
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 5
EAR INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 6
GASTROENTERITIS ROTAVIRUS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
GASTROENTERITIS SALMONELLA (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
LARYNGITIS (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 3
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
MASTOIDITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
ORAL CANDIDIASIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 1 | 2 | 1 | 0 | 0 | 2 | 0 | 6
PYELONEPHRITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
RESPIRATORY SYNCYTIAL VIRUS BRONCHIOLITIS (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
SALMONELLOSIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 3
CONCUSSION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
SKULL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
COW'S MILK INTOLERANCE (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 5
JUVENILE IDIOPATHIC ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
BENIGN INTRACRANIAL HYPERTENSION (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
FEBRILE CONVULSION (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
HYDRONEPHROSIS (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ADENOIDAL HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 3
CHOKING (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
TONSILLAR HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | B_2h3h5_11 (N=252) | B_3h5_11 (N=249) | B_68_11 (N=250) | B_02_2_5 (N=104) | B_02_6_10 (N=300) | BC_35_12 (N=126) | C_35_12 (N=123) | TOTAL (N=1404)
DIARRHOEA (Gastrointestinal disorders) | 96 | 74 | 76 | 12 | 5 | 41 | 49 | 353
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 38 | 0 | 0 | 38
VOMITING (Gastrointestinal disorders) | 69 | 46 | 58 | 8 | 6 | 30 | 31 | 248
CHILLS (General disorders) | 0 | 0 | 0 | 0 | 47 | 0 | 0 | 47
CRYING (General disorders) | 198 | 186 | 157 | 0 | 0 | 105 | 93 | 739
INDURATION (General disorders) | 58 | 23 | 27 | 7 | 6 | 1 | 1 | 123
INJECTION SITE ERYTHEMA (General disorders) | 169 | 160 | 157 | 59 | 180 | 62 | 41 | 828
INJECTION SITE INDURATION (General disorders) | 162 | 118 | 122 | 41 | 124 | 42 | 41 | 650
INJECTION SITE PAIN (General disorders) | 202 | 175 | 168 | 99 | 287 | 114 | 102 | 1147
INJECTION SITE SWELLING (General disorders) | 120 | 76 | 84 | 50 | 146 | 34 | 35 | 545
MALAISE (General disorders) | 0 | 0 | 0 | 0 | 117 | 0 | 0 | 117
PYREXIA (General disorders) | 201 | 192 | 189 | 22 | 47 | 99 | 77 | 827
SWELLING (General disorders) | 26 | 6 | 19 | 6 | 4 | 0 | 0 | 61
BRONCHIOLITIS (Infections and infestations) | 18 | 26 | 13 | 0 | 0 | 6 | 5 | 68
BRONCHITIS (Infections and infestations) | 37 | 36 | 33 | 6 | 7 | 0 | 3 | 122
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 6 | 9 | 18
CONJUNCTIVITIS (Infections and infestations) | 27 | 15 | 17 | 0 | 1 | 2 | 3 | 65
EAR INFECTION (Infections and infestations) | 12 | 9 | 16 | 3 | 0 | 1 | 5 | 46
GASTROENTERITIS (Infections and infestations) | 25 | 23 | 32 | 1 | 3 | 5 | 6 | 95
INFLUENZA (Infections and infestations) | 7 | 4 | 5 | 0 | 3 | 7 | 2 | 28
LARYNGITIS (Infections and infestations) | 12 | 5 | 15 | 0 | 0 | 3 | 0 | 35
NASOPHARYNGITIS (Infections and infestations) | 38 | 31 | 47 | 5 | 5 | 14 | 11 | 151
OTITIS MEDIA (Infections and infestations) | 7 | 4 | 14 | 1 | 2 | 0 | 0 | 28
OTITIS MEDIA ACUTE (Infections and infestations) | 10 | 8 | 14 | 1 | 0 | 12 | 16 | 61
PHARYNGITIS (Infections and infestations) | 11 | 10 | 14 | 2 | 4 | 6 | 10 | 57
RESPIRATORY TRACT INFECTION (Infections and infestations) | 18 | 14 | 28 | 0 | 0 | 3 | 3 | 66
TONSILLITIS (Infections and infestations) | 6 | 3 | 7 | 1 | 2 | 6 | 12 | 37
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 49 | 56 | 54 | 3 | 6 | 59 | 60 | 287
VIRAL INFECTION (Infections and infestations) | 16 | 26 | 14 | 4 | 4 | 11 | 10 | 85
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 35 | 50 | 0 | 0 | 85
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 127 | 0 | 0 | 127
HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 7 | 90 | 0 | 0 | 97
SOMNOLENCE (Nervous system disorders) | 186 | 152 | 144 | 39 | 0 | 93 | 84 | 698
EATING DISORDER (Psychiatric disorders) | 141 | 112 | 121 | 35 | 0 | 67 | 64 | 540
IRRITABILITY (Psychiatric disorders) | 181 | 156 | 153 | 49 | 1 | 95 | 79 | 714
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 3 | 0 | 0 | 8 | 7 | 26
CATARRH (Respiratory, thoracic and mediastinal disorders) | 8 | 14 | 14 | 0 | 2 | 0 | 0 | 38
COUGH (Respiratory, thoracic and mediastinal disorders) | 12 | 6 | 13 | 3 | 5 | 1 | 1 | 41
ERYTHEMA (Skin and subcutaneous tissue disorders) | 20 | 8 | 12 | 6 | 3 | 2 | 0 | 51
RASH (Skin and subcutaneous tissue disorders) | 36 | 28 | 32 | 9 | 21 | 11 | 6 | 143

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreement with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publications of the pooled data (i.e., data from all sites) in the clinical trial.